CLINICAL TRIAL: NCT05914714
Title: Ruxolitinib as Graft-versus-Host Disease Prophylaxis for Allogeneic Stem Cell Transplantation in Aplastic Anemia Patients
Brief Title: Ruxolitinib as GVHD Prophylaxis in AA Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023011-EC-2
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: The Prophylactic Value of Ruxolitinib for aGVHD in HSCT Recipients of AA
MeSH Terms: interventions — ruxolitinib; BID protein, human

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: Ruxolitinib 5 MG BID Oral Tablet

INTERVENTIONS:
Drug: Ruxolitinib 5 MG BID Oral Tablet — ruxolitinib 5mgBID will be administrated at the beginning of the conditioning regimen until 3 months post-transplantation.

SUMMARY:
Our study aimed to determine the prophylactic value of ruxolitinib for aGVHD in HSCT recipients of AA.Ruxolitinib was initiated at the beginning of conditioning regimen at 5 twice daily until 3 months post-transplantation. The cumulative incidence of aGVHD within 6 months after HSCT will be the primary observation item.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed as aplasitic anemia, including V/SAA,CAA and HAAA. (2) Age elder than or equal to 14 years; (3) Informed consent may be signed by themselves. (4) HIV negative, HBV, HCV negative; (5) Informed consent must be signed before the start of the study procedures, and informed consent must be signed by the patient himself or his immediate family. Considering the patient 's condition, if the patient' s signature is unfavorable for disease treatment, the informed consent form should be signed by the legal guardian or the patient 's immediate family member

Exclusion Criteria:

* (1) received a previous allogeneic HSCT; (2) Uncontrolled infection at enrollment; requires mechanical ventilation or is hemodynamically unstable at the time of enrollment; (3) has severe hepatic insufficiency (defined as Child-Pugh Class C; has serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 xthe upper limit of normal (ULN) or serum total bilirubin > 2.5 x ULN.

  (4) has end-stage renal impairment with a creatinine clearance less than 10 mL/min.

  (5) has both moderate hepatic insufficiency AND moderate renal insufficiency; (6) has documented positive results for human immunodeficiency virus antibody (HIVAb), hepatitis C virus antibody (HCV-Ab) with detectable HCV RNA, or hepatitis B surface antigen (HBsAg) within 90 days prior to enrollments; (7) has active solid tumor malignancies with the exception of localized basal cell or squamous cell skin cancer or the condition under treatment (e.g., lymphomas).

  (8) Suffering from mental disorders or other conditions and unable to cooperate with the requirements of study treatment and monitoring; (9) unable or unwilling to sign the consent form; (10) patients with other special conditions assessed as unqualified by the investigator

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
cumulative incidence of aGVHD | 6 months post-HSCT
  cumulative incidence of aGVHD within 6 months post-HSCT

IPD SHARING:
Plan to Share IPD: No